CLINICAL TRIAL: NCT02510235
Title: A Multicenter, Randomized, Double-masked, Controlled, Non-inferiority Study to Evaluate Tolerability, Safety and Efficacy of Lubricin vs Sodium Hyaluronate in Subjects With Moderate Dry Eye.
Brief Title: Tolerability, Safety and Efficacy of Lubricin vs Sodium Hyaluronate Eye Drops in Subjects With Moderate Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LUB0114MD; CIV-15-01-013105 (Other: EudaMed)
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Dry Eye Syndrome; Tear Film Insufficiency
Keywords: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes; Xerophthalmia

STUDY DESIGN:
Intervention Model Description: This was a 4-week randomised (1:1), controlled, double-masked, non-inferiority clinical investigation in subjects with moderate dry eye disease. Subjects with moderate dry eye will be evaluated at screening (from day -14 to day -8), baseline (day 1), week 2 (day 14±2 days), week 4 (day 28±4 days, or early exit) and at week 5 (at least 7 days but not more than 9 days after V4).
  Treatment duration 28 days (4weeks) ± 4 days (maximum total study duration 32 days).
  During the Run-in period of 7 days only a saline solution 0.9%, Nebul®, was allowed to the subject in both eyes four times a day (QID) every 4 h±1 h. No ocular topical treatments were allowed, including artificial tears/lubricants.
  During the follow-up period (7-9 days) only Sodium hyaluronate (Na-HY) 0.13% eye drops monodose supplied by the Investigator will be allowed, to all subjects participating to the study, in both eyes as needed.
Who Masked: Participant, Investigator
Masking Description: The packaging used for the comparator in the present investigation aimed at ensuring a complete masking of the test IMD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lubricin (Experimental): Lubricin 150 µg/ml eye drops. The test investigational device as well as the comparator, was instilled q.i.d.(four times a day), one drop into each eye for 28±4 days. After the end of the treatment period, all the subjects used 0.13% Sodium hyaluronate eye drops (Ocuyal®) q.i.d. for the following 7-9 days.
  Before the start of the treatment (run-in period of 7 days), the subjects were allowed to use NaCl 0.9% ocular solution (Nebul®) q.i.d.
  Interventions: Device: Lubricin
- Sodium Hyaluronate (Active Comparator): Sodium hyaluronate 0.13% eye drops. The comparator, as well as the test investigational device, was instilled q.i.d.(four times a day), one drop into each eye for 28±4 days. After the end of the treatment period, all the subjects used 0.13% Sodium hyaluronate eye drops (Ocuyal®) q.i.d. for the following 7-9 days.
  Before the start of the treatment (run-in period of 7 days), the subjects were allowed to use NaCl 0.9% ocular solution (Nebul®) q.i.d.
  Interventions: Device: Sodium Hyaluronate

INTERVENTIONS:
Device: Lubricin — Lubricin 150 µg/ml eye drops
  Arms: Lubricin
Device: Sodium Hyaluronate — Sodium hyaluronate 0.13% eye drops
  Other Names: Ocuyal®
  Arms: Sodium Hyaluronate

SUMMARY:
The objective of the clinical investigation was to evaluate tolerability, safety and efficacy of the tested medical device, eye drop containing Lubricin 150 µg/mL, as compared with a standard sodium hyaluronate 0.13% eye drop solution in subjects with moderate dry eye disease.

Primary objective:

• Symptom Assessment in Dry Eye (SANDE)

Secondary objectives:

* Treatment-emergent adverse events (TEAEs);
* Visual analogue scale (VAS) for ocular tolerability (foreign body sensation, burning/stinging, itching, pain, stick feeling, blurred vision and photophobia);
* Tear film osmolarity;
* Assessment of best corrected distance visual acuity (BCDVA)
* Slit lamp examination (SLE) to assess the Eyelid - Meibomian glands, Eyelid Erythema, Eyelid Oedema, Lashes, Conjunctiva Erythema, Lens, Iris, Anterior Chamber, Corneal transparency, Corneal neovascularization;
* Tear film break-up time (TFBUT);
* Corneal fluorescein surface staining (scored using the Oxford scale);
* Schirmer-I test (without anaesthesia) values;
* Intraocular Pressure (IOP)

All parameters will be evaluated at screening visit, baseline (day 1), visit 3 (day 14±2) and visit 4 (day 28±4) and at follow-up (final visit) at least 7 days but not more than 9 days after the last treatment.

The results for both the SANDE questionnaire and adverse events are reported at the patient level, without distinguishing between Study Eye and Non-Study Eye. This approach reflects the overall condition and experiences of the patient rather than attributing outcomes to individual eyes.

The Study Eye was identified as the eye with the worst overall tolerability score at Visit 2 (Day 1).

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-masked, controlled, non-inferiority study to evaluate tolerability, safety and efficacy of Lubricin eye drops versus sodium hyaluronate eye drops (Ocuyal®) administered four times a day for 4 weeks and 1 week follow-up in subjects with moderate dry eye.

ELIGIBILITY:
Inclusion Criteria:

To be checked at the screening visit (V1) from day -14 to day -8 days before run-in period and confirmed at baseline visit (V2):

1. Subjects 18 years of age or older.
2. Subjects with moderate dry eye characterized by tear film osmolarity > 312 mOsm
3. Subjects with both VAS for frequency and severity of symptoms, SANDE items, at screening & baseline > 25 mm (SANDE overall score > 25 mm).
4. Subjects with moderate dry eye characterized by at least one eye with signs and symptoms of moderate dry eye (grade 2 or 3 of the 2007 DEWS report)
5. Subjects diagnosed with dry eye from at least 6 months (current use or recommended use of artificial tears/lubricants for the treatment of Dry Eye)
6. Best corrected distance visual acuity (BCDVA) score of ≥ 0.1 decimal units in both eyes at the time of study enrolment.
7. The Informed Consent form approved by the Ethics Committees should be signed by the subject before any study procedures.

Exclusion Criteria:

1. Evidence of an active ocular infection in either eye
2. History or presence of ocular surface disorders not related to dry eye in either eye
3. History or evidence of eyelid abnormality in either eye
4. Use of topical cyclosporine, topical corticosteroids or any other topical medication for the treatment of dry eye in either eye within 30 days of study enrolment
5. History of any ocular surgery (including laser or refractive surgical procedures) in either eye within the 90 days before study enrolment. Ocular surgery will not be allowed during the study treatment period and elective ocular surgery procedures should not be planned during the duration of the follow-up period
6. Presence or history of any ocular or systemic disorder or condition that might significantly hinder the efficacy of the study treatment or its evaluation, could possibly interfere with the interpretation of study results, or could be judged by the investigator to be incompatible with the study visit schedule or conduct of trail procedures (e.g. ocular trauma, progressive or degenerative corneal conditions, uveitis, systemic vasculitis, collagen vascular diseases, poorly controlled diabetes, autoimmune disease, systemic infection.)
7. Known hypersensitivity to one of the components of the test device or the comparator
8. Participation in another clinical study at the same time as the present study or within 90 days of baseline visit
9. History of drug, medication or alcohol abuse or addiction.
10. Females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) are excluded from participation in the study if they meet any one of the following conditions:

    * are currently pregnant or,
    * have a positive result on the urine pregnancy test at the Screening/Baseline Visit or,
    * intend to become pregnant during the study treatment period or,
    * are breast-feeding or,
    * not willing to use highly effective birth control measures, such as: Hormonal contraceptives - oral, implanted, transdermal, or injected and/or mechanical barrier methods - spermicide in conjunction with a barrier such as a condom or diaphragm or IUD during the entire course of and 30 days after the study treatment periods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-03-09; Primary Completion 2015-06-10 (Actual); Study Completion 2015-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Mantelli, MD, Study Director — Dompé farmaceutici
Locations (2):
- Italy (2):
  - Azienda OspedalieroUniversitaria "Policlinico Vittorio Emanuele" Presidio Ospedaliero S.Marta Clinica oculistica, Catania
  - Ambulatorio Studio delle Malattie della Superficie Oculare, Unità Operativa Complessa di Oftalmologia, Azienda Ospedaliero Universitaria di Messina, Messina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was competitive between the study sites and continued until the planned number of randomised patients was achieved. Competitive recruitment was chosen to increase the speed of recruitment and to account for any difference in enrolment rate between study sites.
Pre-assignment Details: Fifty-nine (59) subjects were screened and all of them were eligible for the investigation. Three (3) of the eligible subjects were not randomised and did not receive any treatment. So Fifty-six (56) subjects were randomised 1: 1 to Lubricin or Sodium Hyaluronate and used their assigned IMD at least once.
Groups:
- Lubricin: Lubricin 150 µg/ml eye drops. The test investigational device, as well as the comparator, was instilled q.i.d.(four times a day), one drop into each eye for 28±4 days. After the end of the treatment period, all the subjects used 0.13%Sodium hyaluronate eye drops q.i.d. for the following 7-9 days.
  Before the start of the treatment (run-in period of 7 days), the subjects were allowed to use NaCl 0.9% ocular solution q.i.d.
  Lubricin: Lubricin 150 µg/ml eye drops
- OcuYal®: OcuYal® is sodium hyaluronate 0.13% eye drops. The comparator, as well as the test investigational device, was instilled q.i.d.(four times a day), one drop into each eye for 28±4 days. After the end of the treatment period, all the subjects used 0.13%Sodium hyaluronate eye drops q.i.d. for the following 7-9 days.
  Before the start of the treatment (run-in period of 7 days), the subjects were allowed to use NaCl 0.9% ocular solution q.i.d.
  Sodium Hyaluronate: Sodium hyaluronate 0.13% eye drops
Period: Overall Study
Arm/Group | Lubricin | OcuYal®
Started (Randomised and used their assigned IMD) | 27 | 29
Per-Protocol Population (PP) | 24 | 27
Completed | 26 | 29
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Per Protocol set (PP): all enrolled subjects who fulfilled the investigation protocol requirements in terms of IMD intake (Lubricin or OcuYal®) during the treatment phase and collection of primary efficacy data and with no major deviations that could affect the results. This analysis set was used for the efficacy analysis.
Groups:
- Lubricin: Lubricin 150 µg/ml eye drops. The test investigational device, as well as the comparator, was instilled q.i.d.(four times a day), one drop into each eye for 28±4 days. After the end of the treatment period, all the subjects used 0.13% Sodium hyaluronate eye drops q.i.d. for the following 7-9 days.
  Before the start of the treatment (run-in period of 7 days), the subjects were allowed to use NaCl 0.9% ocular solution q.i.d.
  Lubricin: Lubricin 150 µg/ml eye drops
- Sodium Hyaluronate: Sodium hyaluronate 0.13% eye drops. The comparator, as well as the test investigational device, was instilled q.i.d.(four times a day), one drop into each eye for 28±4 days. After the end of the treatment period, all the subjects used 0.13%Sodium hyaluronate eye drops q.i.d. for the following 7-9 days.
  Before the start of the treatment (run-in period of 7 days), the subjects were allowed to use NaCl 0.9% ocular solution q.i.d.
  Sodium Hyaluronate: Sodium hyaluronate 0.13% eye drops
- Total: Total of all reporting groups
Arm/Group | Lubricin | Sodium Hyaluronate | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Categorical [Count of Participants; unit: Participants] — Population: Fifty-six (56) subjects were randomised and used their assigned IMD at least once.
  Fifty-five (55) of the 56 enrolled subjects completed the investigation per protocol, while one subject prematurely withdrew consent to the participation in the investigation.
  Participants
    PP population: <=18 years | 0 | 0 | 0
    PP population: Between 18 and 65 years | 18 | 17 | 35
    PP population: >=65 years | 6 | 10 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All 56 randomised subjects were included in the safety analysis set. Fifty-five (55) out of 56 safety set subjects were included in the full analysis set (FAS). The per protocol set included 51 subjects.
  years
    PP population | 57.6 (10.6) | 57.7 (12.9) | 57.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All 56 randomised subjects were included in the safety analysis set. Fifty-five (55) out of 56 safety set subjects were included in the full analysis set (FAS). The per protocol set included 51 subjects.
  Participants
    PP population: Female | 18 | 24 | 42
    PP population: Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All 56 randomised subjects were included in the safety analysis set. Fifty-five (55) out of 56 safety set subjects were included in the full analysis set (FAS). The per protocol set included 51 subjects.
  Participants
    PP population: American Indian or Alaska Native | 0 | 0 | 0
    PP population: Asian | 0 | 0 | 0
    PP population: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    PP population: Black or African American | 0 | 0 | 0
    PP population: White | 24 | 27 | 51
    PP population: More than one race | 0 | 0 | 0
    PP population: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 24 | 27 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (V2) in Frequency and Severity of Dry Eye Symptoms (SANDE) Questionnaire Scores at Day 28±4 (End of Treatment)
Description: The SANDE (Symptom Assessment in Dry Eye) questionnaire was used to evaluate both dry eye frequency and severity using a 100 mm VAS line, representing ocular dryness and/or irritation at subject's level, according to their own perception, irrespective of the eye being or not the study eye, as per study Protocol. SANDE scores ranged from 0 (best condition) to 100 (worst condition) for both severity and frequency. The VAS score was determined - in millimeters - by measuring from the left-hand end to the marked point on the VAS line. SANDE OVERALL VAS score was calculated considering the mean and the SD of the "Change from Baseline" values at Day 14±2, Day 28±4 and Day 31-41, both for frequency and severity, and then calculated as square-root of the product of the two item score. Results are reported at the patient level, rather than focusing on a single eye, as the SANDE score assesses overall dry eye symptoms rather than eye-specific effects, as per study protocol.
Time Frame: Visit 3 - Day 14±2, Visit 4 - Day 28±4, Visit 5 - Final visit/Follow up - Day 31- 41
Population: The Per Protocol set (PP) population included all enrolled subjects who fulfilled the investigation protocol requirements in terms of IMD intake (Lubricin or OcuYal®) during the treatment phase and collection of primary efficacy data and with no major deviations that could affect the results. This analysis set was used for the efficacy analysis.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Lubricin PP: Lubricin 150 µg/ml eye drops. The test investigational device as well as the comparator, was instilled q.i.d.(four times a day), one drop into each eye for 28±4 days. After the end of the treatment period, all the subjects used 0.13% Sodium hyaluronate eye drops q.i.d. for the following 7-9 days.
  Before the start of the treatment (run-in period of 7 days), the subjects were allowed to use NaCl 0.9% ocular solution q.i.d.
  Lubricin: Lubricin 150 µg/ml eye drops
- Sodium Hyaluronate PP: Sodium hyaluronate 0.13% eye drops. The comparator, as well as the test investigational device, was instilled q.i.d.(four times a day), one drop into each eye for 28±4 days. After the end of the treatment period, all the subjects used 0.13%Sodium hyaluronate eye drops q.i.d. for the following 7-9 days.
  Before the start of the treatment (run-in period of 7 days), the subjects were allowed to use NaCl 0.9% ocular solution q.i.d.
  Sodium Hyaluronate: Sodium hyaluronate 0.13% eye drops
Arm/Group | Lubricin PP | Sodium Hyaluronate PP
Number analyzed (Participants) | 24 | 27
mm
  Day 14±2 - Frequency | -11.9 (8.6) | -16.6 (14.9)
  Day 28±4 -Frequency | -25.0 (12.2) | -26.5 (18.0)
  Day 31-41 - Frequency | -27.8 (14.5) | -30.9 (19.2)
  Day 14±2 - Severity | -10.6 (6.0) | -13.7 (12.8)
  Day 28±4 - Severity | -22.2 (14.1) | -21.8 (14.1)
  Day 31-41 - Severity | -25.6 (16.6) | -25.4 (14.5)
  Day 14±2 - Overall Score | -11.2 (6.9) | -15.3 (13.6)
  Day 28±4 - Overall score | -23.5 (11.9) | -24.2 (15.7)
  Day 31-41 - Overall Score | -26.6 (13.4) | -28.3 (16.5)
Statistical Analysis 1: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Values at Day 28 ± 4 (end of treatment) for the SANDE overall VAS score were compared between treatment groups using a Student's t-test for unpaired data; Test type: Non-Inferiority — To declare non-inferiority between treatments, a change in the SANDE overall score of 12 mm was required, with an estimated standard deviation of 13 (approximately 70% of the mean at 28 ± 4 days after treatment). The left inferior limits of confidence interval were determined and compared with the non-inferiority limit defined in the testing hypothesis. Testing Hypothesis: H0: meanHyaluronic - meanLubricin ≤ - 12 / H1: meanHyaluronic - meanLubricin > - 12; Student t-test for unpaired data; Mean Difference (Final Values) = 1.50, 95% CI 1-sided [lower limit -8.87]

2. Secondary Outcome: Treatment-emergent Adverse Events (TEAEs), Including Adverse Device Effects (ADEs)
Description: Occurrence of Treatment-emergent adverse events (TEAEs), including adverse device effects (ADEs) assessed throughout the study after the first IMD administration.
Time Frame: From Visit 2 (Day 1)" i.e., the day of the first IMD administration to Visit 5 - Final visit/Follow up - Day 31- 41
Population: The Safety Population (SAF) included all subjects who received at least one dose of the IMDs (Lubricin or Sodium Hyaluronate-OcuYal®).
Measure: Number; unit: Number of adverse events
Groups:
- Lubricin SAF: Lubricin 150 µg/ml eye drops. The test investigational device as well as the comparator, was instilled q.i.d.(four times a day), one drop into each eye for 28±4 days. After the end of the treatment period, all the subjects used 0.13% Sodium hyaluronate eye drops q.i.d. for the following 7-9 days.
  Before the start of the treatment (run-in period of 7 days), the subjects were allowed to use NaCl 0.9% ocular solution q.i.d.
  Lubricin: Lubricin 150 µg/ml eye drops
- Sodium Hyaluronate SAF: Sodium hyaluronate 0.13% eye drops. The comparator, as well as the test investigational device, was instilled q.i.d.(four times a day), one drop into each eye for 28±4 days. After the end of the treatment period, all the subjects used 0.13%Sodium hyaluronate eye drops q.i.d. for the following 7-9 days.
  Before the start of the treatment (run-in period of 7 days), the subjects were allowed to use NaCl 0.9% ocular solution q.i.d.
  Sodium Hyaluronate: Sodium hyaluronate 0.13% eye drops
Arm/Group | Lubricin SAF | Sodium Hyaluronate SAF
Number analyzed (Participants) | 27 | 29
Number of adverse events
  All TEAEs | 4 | 6
  TEAEs - Related to Treatment | 4 | 0
  TEAEs - Not Related to Treatment | 0 | 6
  TEAEs - Unknown | 0 | 5
  TEAEs - Mild | 0 | 0
  TEAEs - Moderate | 4 | 1
  TEAEs - Severe | 0 | 0
  All serious TEAEs | 0 | 0
  TEAEs - Leading to discontinuation | 4 | 0

3. Secondary Outcome: Changes From Baseline (Visit 2, Day 1) in Ocular Tolerability Using a Visual Analogue Scale (VAS)
Description: A global ocular tolerability score was determined using a 100 mm Visual Analogue Scale (VAS) on which 0 meant no symptoms and 100 meant the worst possible discomfort. This evaluation was to be performed before any ophthalmic assessment at each scheduled visit. Specific ocular symptoms measured with the VAS included: foreign body sensation, burning/stinging, itching, pain, sticky feeling, blurred vision, photophobia. The patients evaluated their symptoms using the VAS giving the value they were feeling from none to an extreme value. The VAS scale was a straight horizontal line of fixed length (100 mm). The ends were defined as extreme limits of the parameter.
Time Frame: Visit 3 - Day 14±2, Visit 4 - Day 28±4, Visit 5 - Final visit/Follow up - Day 31- 41
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Lubricin PP: Lubricin 150 µg/ml eye drops. The test investigational device as well as the comparator, was instilled q.i.d.(four times a day), one drop into each eye for 28±4 days. After the end of the treatment period, all the subjects used 0.13% Sodium hyaluronate eye drops (Ocuyal®) q.i.d. for the following 7-9 days.
  Before the start of the treatment (run-in period of 7 days), the subjects were allowed to use NaCl 0.9% ocular solution (Nebul®) q.i.d.
  Lubricin: Lubricin 150 µg/ml eye drops
- Sodium Hyaluronate PP: Sodium hyaluronate 0.13% eye drops. The comparator, as well as the test investigational device, was instilled q.i.d.(four times a day), one drop into each eye for 28±4 days. After the end of the treatment period, all the subjects used 0.13% Sodium hyaluronate eye drops (Ocuyal®) q.i.d. for the following 7-9 days.
  Before the start of the treatment (run-in period of 7 days), the subjects were allowed to use NaCl 0.9% ocular solution (Nebul®) q.i.d.
  Sodium Hyaluronate: Sodium hyaluronate 0.13% eye drops
Arm/Group | Lubricin PP | Sodium Hyaluronate PP
Number analyzed (Participants) | 24 | 27
mm
  Foreign Body sensation - Study eye -Day 14±2 | -12.6 (11.4) | -16.2 (15.4)
  Foreign Body sensation - Non Study eye -Day 14±2 | -9.4 (10.8) | -11.7 (10.4)
  Burning /Stinging - Study eye - Day 14±2 | -15.9 (13.5) | -15.7 (17.2)
  Burning /Stinging - Non Study eye - Day 14±2 | -8.9 (12.1) | -8.6 (10.1)
  Itching - Study eye - Day 14±2 | -15.7 (12.7) | -10.9 (15.0)
  Itching - Non Study eye - Day 14±2 | -10.9 (15.7) | -8.9 (12.6)
  Pain - Study eye - Day 14±2 | -13.7 (13.0) | -14.2 (17.3)
  Pain - Non Study eye - Day 14±2 | -8.2 (12.8) | -10.7 (11.0)
  Sticky feeling- Study eye - Day 14±2 | -13.5 (12.5) | -5.6 (15.0)
  Sticky feeling- Non Study eye - Day 14±2 | -11.2 (9.8) | -5.7 (12.2)
  Blurred vision- Study eye - Day 14±2 | -11.3 (16.1) | -12.0 (15.3)
  Blurred vision- Non Study eye - Day 14±2 | -9.1 (14.5) | -5.7 (12.0)
  Photophobia - Study eye - Day 14±2 | -19.5 (17.3) | -18.5 (17.5)
  Photophobia - Non Study eye - Day 14±2 | -11.7 (13.4) | -19.5 (20.9)
  Total score - Study eye - Day 14±2 | -102.2 (64.2) | -93.2 (74.3)
  Total score - Non Study eye - Day 14±2 | -69.5 (48.9) | -70.9 (56.3)
  Foreign Body sensation - Study eye -Day 28±4 | -25.0 (17.6) | -26.7 (19.8)
  Foreign Body sensation - Non Study eye -Day 28±4 | -17.0 (17.3) | -21.8 (12.1)
  Burning /Stinging - Study eye - Day 28±4 | -27.6 (18.36) | -23.0 (20.0)
  Burning /Stinging - Non Study eye - Day 28±4 | -14.6 (16.3) | -12.3 (15.6)
  Itching - Study eye - Day 28±4 | -27.6 (18.5) | -18.5 (17.3)
  Itching - Non Study eye - Day 28±4 | -19.3 (16.8) | -15.1 (16.2)
  Pain - Study eye - Day 28±4 | -24.1 (18.4) | -20.1 (18.4)
  Pain - Non Study eye - Day 28±4 | -15.0 (18.8) | -14.5 (15.3)
  Sticky feeling- Study eye - Day 28±4 | -21.9 (18.6) | -13.1 (21.5)
  Sticky feeling - Non Study eye - Day 28±4 | -17.6 (19.4) | -9.2 (18.0)
  Blurred vision - Study eye - Day 28±4 | -14.0 (19.4) | -15.6 (24.5)
  Blurred vision - Non Study eye - Day 28±4 | -13.4 (18.6) | -8.8 (19.0)
  Photophobia - Study eye - Day 28±4 | -28.8 (25.1) | -26.1 (23.4)
  Photophobia - Non Study eye - Day 28±4 | -17.1 (27.1) | -23.3 (26.2)
  Total score - Study eye - Day 28±4 | -168.9 (82.8) | -143.1 (107.5)
  Total score - Non Study eye - Day 28±4 | -114.1 (74.3) | -105.0 (75.9)
  Foreign Body sensation - Study eye - Day 31-41 | -28.3 (21.8) | -28.1 (18.2)
  Foreign Body sensation - Non study eye - Day 31-41 | -19.7 (15.8) | -18.4 (14.2)
  Burning/Stinging -Study eye -Day 31-41 | -30.5 (23.5) | -23.6 (20.2)
  Burning/Stinging - Non study eye - Day 31-41 | -11.1 (19.2) | -14.1 (18.6)
  Itching - Study eye - Day 31-41 | -28.6 (22.9) | -19.1 (21.4)
  Itching - Non study eye - Day 31-41 | -18.9 (17.5) | -15.7 (21.4)
  Pain - Study eye - Day 31-41 | -26.9 (20.1) | -20.7 (18.0)
  Pain - Non study eye - Day 31-41 | -12.0 (21.7) | -18.6 (19.4)
  Sticky feeling - Study eye - Day 31-41 | -20.5 (23.1) | -13.3 (19.4)
  Sticky feeling - Non study eye - Day 31-41 | -21.4 (21.8) | -5.2 (16.3)
  Blurred vision - Study eye - Day 31-41 | -14.6 (19.4) | -15.3 (23.9)
  Blurred vision - Non study eye - Day 31-41 | -10.9 (19.8) | -9.8 (18.7)
  Photophobia - Study eye - Day 31-41 | -25.3 (25.1) | -24.9 (26.0)
  Photophobia - Non study eye - Day 31-41 | -17.6 (27.5) | -19.9 (26.6)
  Total score - Study eye - Day 31-41 | -174.8 (96.0) | -145.1 (102.2)
  Total score - Non study eye - Day 31-41 | -11.5 (86.2) | -101.4 (95.8)
Statistical Analysis 1: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Foreign Body Sensation in the Study Eye was analyzed using a repeated measures ANOVA, which evaluates changes from baseline across all time points in a single analysis. This method provides one overall value for comparison, as it incorporates all time points into a unified analysis. Consequently, the reported value represents the global outcome across time points, consistent with the repeated measures ANOVA methodology; Test type: Superiority; p = 0.8226, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-7.66 to 6.11]
Statistical Analysis 2: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Burning/Stinging in Study eye was analyzed using a repeated measures ANOVA, which evaluates changes from baseline across all time points in a single analysis. This method provides one overall value for comparison, as it incorporates all time points into a unified analysis. Consequently, the reported value represents the global outcome across time points, consistent with the repeated measures ANOVA methodology; Test type: Superiority; p = 0.3178, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = 3.16, 95% CI 2-sided [-3.13 to 9.44]
Statistical Analysis 3: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Itching in Study eye was analyzed using a repeated measures ANOVA, which evaluates changes from baseline across all time points in a single analysis. This method provides one overall value for comparison, as it incorporates all time points into a unified analysis. Consequently, the reported value represents the global outcome across time points, consistent with the repeated measures ANOVA methodology; Test type: Superiority; p = 0.0085, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = 6.52, 95% CI 2-sided [1.74 to 11.30]
Statistical Analysis 4: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Pain in Study eye was analyzed using a repeated measures ANOVA, which evaluates changes from baseline across all time points in a single analysis. This method provides one overall value for comparison, as it incorporates all time points into a unified analysis. Consequently, the reported value represents the global outcome across time points, consistent with the repeated measures ANOVA methodology; Test type: Superiority; p = 0.3124, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = 3.41, 95% CI 2-sided [-3.31 to 10.13]
Statistical Analysis 5: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Sticky feeling in Study eye was analyzed using a repeated measures ANOVA, which evaluates changes from baseline across all time points in a single analysis. This method provides one overall value for comparison, as it incorporates all time points into a unified analysis. Consequently, the reported value represents the global outcome across time points, consistent with the repeated measures ANOVA methodology; Test type: Superiority; p = 0.0377, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = 6.76, 95% CI 2-sided [0.40 to 13.12]
Statistical Analysis 6: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Blurred vision in Study eye was analyzed using a repeated measures ANOVA, which evaluates changes from baseline across all time points in a single analysis. This method provides one overall value for comparison, as it incorporates all time points into a unified analysis. Consequently, the reported value represents the global outcome across time points, consistent with the repeated measures ANOVA methodology; Test type: Superiority; p = 0.5321, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = 2.10, 95% CI 2-sided [-4.62 to 8.83]
Statistical Analysis 7: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Photophobia in Study eye was analyzed using a repeated measures ANOVA, which evaluates changes from baseline across all time points in a single analysis. This method provides one overall value for comparison, as it incorporates all time points into a unified analysis. Consequently, the reported value represents the global outcome across time points, consistent with the repeated measures ANOVA methodology; Test type: Superiority; p = 0.5790, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = 2.32, 95% CI 2-sided [-6.04 to 10.68]
Statistical Analysis 8: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Total ocular tolerability score in Study eye was analyzed using a repeated measures ANOVA, which evaluates changes from baseline across all time points in a single analysis. This method provides one overall value for comparison, as it incorporates all time points into a unified analysis. Consequently, the reported value represents the global outcome across time points, consistent with the repeated measures ANOVA methodology; Test type: Superiority; p = 0.3383, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = 16.13, 95% CI 2-sided [-17.41 to 49.68]

4. Secondary Outcome: Change From Baseline in Tear Film Osmolarity
Description: Tear film osmolarity as a marker of tear film solute content was performed with a TearLab Osmolarity System. The concentration of the tears was assessed in both eyes before the instillation of any dilating or anaesthetic drops. The tear fluid was collected onto the bottom tip of the test card by passive capillary action. After a successful tear collection, the Pen was docked into the Reader, which showed the quantitative tear film osmolarity result in mOsm/L on the liquid crystal display. Normal Patients: 275-316 mOsms/L (mean 302 mOsms/L), Dry Eye Disease Patients: > 316 mOsms/L. The higher the score the worst the outcome.
Time Frame: Visit 3 - Day 14±2, Visit 4 - Day 28±4, Visit 5 - Final visit/Follow up - Day 31- 41
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mOsm /L
Arm/Group | Lubricin PP | Sodium Hyaluronate PP
Number analyzed (Participants) | 24 | 27
mOsm /L
  Day 14±2 - Study eye | -9.6 (15.0) | -12.7 (11.8)
  Day 14±2 - Non Study eye | -10.3 (8.4) | -12.1 (11.5)
  Day 28±4 - Study eye | -7.0 (24.4) | -12.4 (11.3)
  Day 28±4 - Non study eye | -10.8 (11.4) | -12.7 (13.0)
  Day 31-41 - Study eye | -7.6 (14.4) | -9.2 (10.2)
  Day 31-41 - Non study eye | -7.8 (8.0) | -11.2 (11.5)
Statistical Analysis 1: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Study Eye analytic statistic is presented. The Statistical Analysis section reports results from a repeated measures ANOVA, which analyzes changes from baseline across all time points in a single unified analysis. This approach provides one overall comparison value by incorporating all time points. Consequently, the reported value represents the global outcome, consistently with repeated measures ANOVA methodology; Test type: Superiority; p = 0.6484, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-5.07 to 3.19]

5. Secondary Outcome: Change From Baseline in Best Corrected Distance Visual Acuity (BCDVA) - ETDRS Score
Description: Best corrected visual acuity (BCDVA) was determined by careful refraction according to the standard protocol for refraction. Chart 1 was used for testing the VA of the right eye; Chart 2 for the left eye; and Chart R for refraction only. Retroilluminated standard Early Treatment of Diabetic Retinopathy Study (ETDRS) charts were used. They had 5 Sloan letters on each line of equal difficulty, and there was a geometric progression in letter size from line to line. VAS awarded one point for every letter correctly guessed. A distance of 4 meters was required between the subject's eyes and the VA chart. When a subject cannot read at least 20 letters on the chart at 4 meters, the subject was tested at 1 meter. If 20 or more letters were read at 4 meters, the VAS for that eye was recorded as the number of letters correct at 4 meters plus 30. Otherwise, the VAS was the number of letters read correctly at 1 meter plus the number read at 4 meters. The higher the score the better the outcome.
Time Frame: Visit 3 - Day 14±2, Visit 4 - Day 28±4, Visit 5 - Final visit/Follow up - Day 31- 41
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lubricin PP | Sodium Hyaluronate PP
Number analyzed (Participants) | 24 | 27
score on a scale
  Day 14±2 - Study eye | 0.0 (1.2) | -0.1 (1.0)
  Day 14±2 -Non study eye | -0.2 (0.8) | -0.3 (1.3)
  Day 28±4 - Study eye | 0.0 (1.6) | -0.3 (1.5)
  Day 28±4 - Non study eye | 0.0 (1.2) | -0.4 (1.8)
  Day 31-41 - Study eye | 0.1 (1.8) | -0.2 (1.9)
  Day 31-41 - Non study eye | -0.3 (1.3) | -0.5 (1.8)
Statistical Analysis 1: Comparison: Lubricin PP vs Sodium Hyaluronate PP; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.7408, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.71 to 0.51]

6. Secondary Outcome: Change From Baseline in Permanence of Lubricin on the Ocular Surface - Tear Film Break-up Time (TFBUT)
Description: TFBUT was measured by determining the time to tear break-up. The TFBUT test was performed after instillation of 5 μl of 2% preservative-free sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye. With the aid of a slit lamp at 10X magnification using cobalt blue illumination, the examiner monitored the integrity of the tear film, noting the time it took to form lacunae (clear spaces in the tear film) from the time that the eye was opened after the last blink. This measurement was performed within 10 seconds maximum. The TFBUT was measured twice during the first minute after the instillation of the fluorescein. If the 2 readings differed by more than 2 seconds, a third reading was taken. The TFBUT value was the average of the 2 or 3 measurements. Generally, a TFBUT value of 10-35 seconds was considered normal. A value of less than 10 seconds was usually suspicious and may indicate tear film instability. The higher the value, the better the outcome.
Time Frame: Visit 3 - Day 14±2, Visit 4 - Day 28±4, Visit 5 - Final visit/Follow up - Day 31- 41
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Lubricin PP | Sodium Hyaluronate PP
Number analyzed (Participants) | 24 | 27
seconds
  Day 14±2 - Study eye | 1.0 (2.0) | 1.1 (2.5)
  Day 14±2 - Non study eye | 0.6 (2.7) | 1.6 (2.6)
  Day 28±4 - Study eye | 1.3 (2.1) | 1.9 (2.7)
  Day 28±4 - Non study eye | 0.3 (2.8) | 2.5 (2.8)
  Day 31-41 - Study eye | 0.5 (1.8) | 1.0 (1.8)
  Day 31-41 - Non study eye | 0.5 (2.5) | 1.4 (2.0)
Statistical Analysis 1: Comparison: Lubricin PP vs Sodium Hyaluronate PP; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.8596, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.78 to 0.87]

7. Secondary Outcome: Change From Baseline in Slit Lamp Examination (SLE) Values
Description: The Slit Lamp Examination was used to examine the structures of the eye (eyelids, lashes, conjunctiva, cornea, lens, iris and anterior chamber) according to different scales: Eyelid - Meibomian glands (from 0-none to 3-severe), Eyelid - Erythema (from 0-none to 4-very severe), Eyelid - Oedema (from 0-none to 4-very severe), Lashes (0-normal 1-abnormal), Conjunctiva - Erythema (from 0-none to 3-severe), Conjunctiva - Oedema (from 0-none to 4-very severe), Lens (to 0-no opacification to 3-severe opacification), Iris (0-normal 1-abnormal), Anterior chamber inflammation (from 0-none to 3-severe), Cornea transparency (from 0-completely transparent to 4-complete cornea opacity), Cornea neovascularization (0-absence of vascularization to 4- neovascularization between 270° and 360°). The higher the score the worse the outcome. There was not a total score.
Time Frame: Visit 3 - Day 14±2, Visit 4 - Day 28±4, Visit 5 - Final visit/Follow up - Day 31- 41
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lubricin PP | Sodium Hyaluronate PP
Number analyzed (Participants) | 24 | 27
score on a scale
  Eyelid - Meibomian gland - Study eye - Day 14±2 | -0.5 (0.6) | -0.4 (0.5)
  Eyelid - Meibomian gland - Non study eye - Day 14±2 | -0.5 (0.6) | -0.4 (0.6)
  Eyelid - Erythema - Study eye - Day 14±2 | -0.3 (0.6) | -0.4 (0.7)
  Eyelid - Erythema - Non study eye - Day 14±2 | -0.2 (0.6) | -0.4 (0.7)
  Eyelid - Oedema - Study eye - Day 14±2 | -0.2 (0.5) | -0.1 (0.6)
  Eyelid - Oedema - Non study eye - Day 14±2 | -0.2 (0.4) | -0.1 (0.5)
  Lashes - Study eye - Day 14±2 | 0.0 (0.0) | 0.0 (0.0)
  Lashes - Non study eye - Day 14±2 | 0.0 (0.0) | 0.0 (0.0)
  Conjunctiva - Erythema - Study eye - Day 14±2 | -0.4 (0.6) | -0.4 (0.7)
  Conjunctiva - Erythema - Non study eye - Day 14±2 | -0.3 (0.6) | -0.4 (0.8)
  Conjunctiva - Oedema - Study eye - Day 14±2 | 0.0 (0.5) | -0.1 (0.7)
  Conjunctiva - Oedema - Non study eye - Day 14±2 | -0.1 (0.5) | -0.1 (0.6)
  Lens - Study eye - Day 14±2 | 0.0 (0.2) | 0.0 (0.3)
  Lens - Non study eye - Day 14±2 | 0.0 (0.2) | 0.0 (0.2)
  Iris - Study eye - Day 14±2 | 0.0 (0.0) | 0.0 (0.0)
  Iris - Non study eye - Day 14±2 | 0.0 (0.0) | 0.0 (0.0)
  Anterior chamber inflammation - Study eye - Day 14±2 | 0.0 (0.0) | 0.0 (0.0)
  Anterior chamber inflammation - Non study eye - Day 14±2 | 0.0 (0.0) | 0.0 (0.0)
  Cornea transparency - Study eye - Day 14±2 | 0.0 (0.2) | 0.0 (0.2)
  Cornea transparency - Non study eye - Day 14±2 | 0.0 (0.2) | 0.0 (0.2)
  Cornea neovascularisation - Study eye - Day 14±2 | 0.0 (0.0) | 0.0 (0.0)
  Cornea neovascularisation - Non study eye - Day 14±2 | 0.0 (0.0) | 0.0 (0.0)
  Eyelid - Meibomian gland - Study eye - Day 28±4 | -0.5 (0.7) | -0.7 (0.7)
  Eyelid - Meibomian gland - Non study eye -Day 28±4 | -0.5 (0.8) | -0.6 (0.7)
  Eyelid - erythema - Study eye - Day 28±4 | -0.5 (0.7) | -0.4 (0.8)
  Eyelid - erythema - Non study eye - Day 28±4 | -0.5 (0.9) | -0.4 (0.8)
  Eyelid - Oedema - Study eye - Day 28±4 | -0.3 (0.8) | -0.3 (0.8)
  Eyelid - Oedema - Non study eye - Day 28±4 | -0.3 (0.7) | -0.2 (0.7)
  Lashes - Study eye - Day 28±4 | 0.0 (0.0) | 0.0 (0.0)
  Lashes - Non study eye - Day 28±4 | 0.0 (0.0) | 0.0 (0.0)
  Conjunctiva - erythema - Study eye - Day 28±4 | -0.6 (0.8) | -0.6 (0.8)
  Conjunctiva - erythema - Non study eye - Day 28±4 | -0.4 (0.9) | -0.5 (0.9)
  Conjunctiva - Oedema - Study eye - Day 28±4 | -0.2 (0.7) | 0.0 (0.8)
  Conjunctiva - Oedema - Non study eye - Day 28±4 | 0.0 (0.7) | -0.1 (0.8)
  Lens - Study eye - Day 28±4 | 0.0 (0.2) | 0.0 (0.3)
  Lens - Non study eye - Day 28±4 | 0.0 (0.2) | 0.0 (0.2)
  Iris - Study eye - Day 28±4 | 0.0 (0.0) | 0.0 (0.0)
  Iris - Non study eye - Day 28±4 | 0.0 (0.0) | 0.0 (0.0)
  Anterior chamber inflammation - Study eye - Day 28±4 | 0.0 (0.0) | 0.0 (0.0)
  Anterior chamber inflammation - Non study eye - Day 28±4 | 0.0 (0.0) | 0.0 (0.0)
  Cornea tranparency - Study eye - Day 28±4 | 0.0 (0.2) | 0.0 (0.2)
  Cornea tranparency - Non study eye - Day 28±4 | 0.0 (0.2) | 0.0 (0.2)
  Cornea neovascularization - Study eye - Day 28±4 | 0.0 (0.0) | 0.0 (0.0)
  Cornea neovascularization - Non study eye - Day 28±4 | 0.0 (0.0) | 0.0 (0.0)
  Eyelid - Meibomian gland - Study eye - Day 31-41 | -0.6 (0.8) | -0.9 (0.8)
  Eyelid - Meibomian gland - Non study eye - Day 31-41 | -0.7 (0.9) | -0.7 (0.8)
  Eyelid - erythema - Study eye - Day 31-41 | -0.6 (0.7) | -0.6 (0.8)
  Eyelid - erythema - Non study eye - Day 31-41 | -0.6 (0.9) | -0.4 (0.8)
  Eyelid - Oedema - Study eye - Day 31-41 | -0.4 (0.7) | 0.0 (0.6)
  Eyelid - Oedema - Non study eye - Day 31-41 | -0.3 (0.9) | 0.0 (0.6)
  Lashes - Study eye - Day 31-41 | 0.0 (0.0) | 0.0 (0.0)
  Lashes - Non study eye - Day 31-41 | 0.0 (0.0) | 0.0 (0.0)
  Conjunctiva - erythema - Study eye - Day 31-41 | -0.8 (1.0) | -0.4 (1.0)
  Conjunctiva - erythema - Non study eye - Day 31-41 | -0.5 (1.0) | -0.4 (0.9)
  Conjunctiva - Oedema - Study eye - Day 31-41 | -0.1 (0.9) | 0.0 (0.9)
  Conjunctiva - Oedema - Non study eye - Day 31-41 | 0.0 (0.8) | -0.1 (0.9)
  Lens - Study eye - Day 31-41 | 0.0 (0.2) | 0.0 (0.4)
  Lens - Non study eye - Day 31-41 | 0.0 (0.2) | -0.1 (0.3)
  Iris - Study eye - Day 31-41 | 0.0 (0.0) | 0.0 (0.0)
  Iris - Non study eye - Day 31-41 | 0.0 (0.0) | 0.0 (0.0)
  Anterior chamber inflammation - Study eye - Day 31-41 | 0.0 (0.0) | 0.0 (0.0)
  Anterior chamber inflammation - Non study eye - Day 31-41 | 0.0 (0.0) | 0.0 (0.0)
  Cornea transparency - Study eye - Day 31-41 | 0.0 (0.0) | 0.0 (0.2)
  Cornea transparency - Non study eye - Day 31-41 | 0.0 (0.0) | 0.0 (0.2)
  Cornea neovascularization - Study eye - Day 31-41 | 0.0 (0.0) | 0.0 (0.0)
  Cornea neovascularization - Non study eye - Day 31-41 | 0.0 (0.0) | 0.0 (0.0)
Statistical Analysis 1: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Eyelid - Meibomian glands in Study eye analytic statistic is presented. The Statistical Analysis section reports results from a repeated measures ANOVA, which analyzes changes from baseline across all time points in a single unified analysis. This approach provides one overall comparison value by incorporating all time points. Consequently, the reported value represents the global outcome, consistently with repeated measures ANOVA methodology; Test type: Superiority; p = 0.7891, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.16 to 0.20]
Statistical Analysis 2: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Eyelid - Erythema in Study eye analytic statistic is presented. The Statistical Analysis section reports results from a repeated measures ANOVA, which analyzes changes from baseline across all time points in a single unified analysis. This approach provides one overall comparison value by incorporating all time points. Consequently, the reported value represents the global outcome, consistently with repeated measures ANOVA methodology; Test type: Superiority; p = 0.6075, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.24 to 0.14]
Statistical Analysis 3: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Eyelid - Oedema in Study eye analytic statistic is presented.The Statistical Analysis section reports results from a repeated measures ANOVA, which analyzes changes from baseline across all time points in a single unified analysis. This approach provides one overall comparison value by incorporating all time points. Consequently, the reported value represents the global outcome, consistently with repeated measures ANOVA methodology; Test type: Superiority; p = 0.6639, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.14 to 0.21]
Statistical Analysis 4: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Conjunctiva - Erythema in Study eye analytic statistic is presented.The Statistical Analysis section reports results from a repeated measures ANOVA, which analyzes changes from baseline across all time points in a single unified analysis. This approach provides one overall comparison value by incorporating all time points. Consequently, the reported value is not duplicated or triplicated, reflecting the global outcome consistent with repeated measures ANOVA methodology; Test type: Superiority; p = 0.3482, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.10 to 0.29]
Statistical Analysis 5: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Conjunctiva - Oedema in Study eye analytic statistic is presented.The Statistical Analysis section reports results from a repeated measures ANOVA, which analyzes changes from baseline (Visit 2 - Day 1) across all time points in a single unified analysis. This approach provides one overall comparison value by incorporating all time points. Consequently, the reported value represents the global outcome, consistently with repeated measures ANOVA methodology; Test type: Superiority; p = 0.2422, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.34 to 0.09]
Statistical Analysis 6: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Lens in Study eye analytic statistic is presented.The Statistical Analysis section reports results from a repeated measures ANOVA, which analyzes changes from baseline across all time points in a single unified analysis. This approach provides one overall comparison value by incorporating all time points. Consequently, the reported value represents the global outcome, consistently with repeated measures ANOVA methodology; Test type: Superiority; p = 0.8645, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.11 to 0.14]
Statistical Analysis 7: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Cornea transparency in Study eye analytic statistic is presented.The Statistical Analysis section reports results from a repeated measures ANOVA, which analyzes changes from baseline across all time points in a single unified analysis. This approach provides one overall comparison value by incorporating all time points. Consequently, the reported value represents the global outcome, consistently with repeated measures ANOVA methodology; Test type: Superiority; p = 0.3790, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.11 to 0.04]

8. Secondary Outcome: Change From Baseline in Corneal Fluorescein Surface Staining (Oxford Score)
Description: The corneal fluorescein staining was graded by using the Oxford scheme to assess cornea and conjunctiva epithelium damage. The Oxford grading scale divides corneal staining into six groups according to severity from 0 (absent) to 5 (severe). The examiner compared the overall appearance of the patient's corneal staining with a reference figure, simulating the pattern of staining encountered in dry eye disease. No attempt was made to count the dots or to assess the position or confluence of the dots. The examiner selected the appropriate grade that best represented the state of corneal staining. The grading system recommended by NEI divides the cornea into five zones (central, superior, temporal, nasal, and inferior) and for each zone, the severity of corneal fluorescein staining is graded on a scale from 0 to 3 based on reference figures. Therefore, the maximum score (worst outcome) was 15, the minimum (best outcome) was 0.
Time Frame: Visit 3 - Day 14±2, Visit 4 - Day 28±4, Visit 5 - Final visit/Follow up - Day 31- 41
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lubricin PP | Sodium Hyaluronate PP
Number analyzed (Participants) | 24 | 27
score on a scale
  Day 14±2 - Study eye | -0.3 (0.4) | -0.4 (0.6)
  Day 14±2 - Non study eye | -0.3 (0.5) | -0.5 (0.8)
  Day 28±4 - Study eye | -0.9 (0.9) | -0.8 (0.9)
  Day 28±4 - Non study eye | -0.7 (0.6) | -0.7 (0.9)
  Day 31-41 - Study eye | -1.0 (0.9) | -1.0 (0.9)
  Day 31-41 - Non study eye | -1.0 (0.9) | -0.7 (1.0)
Statistical Analysis 1: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Study eye analytic statistic is presented.The Statistical Analysis section reports results from a repeated measures ANOVA, which analyzes changes from baseline across all time points in a single unified analysis. This approach provides one overall comparison value by incorporating all time points. Consequently, the reported value represents the global outcome, consistently with repeated measures ANOVA methodology; Test type: Superiority; p = 0.8363, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.26 to 0.21]

9. Secondary Outcome: Change From Baseline in Schirmer's Test Type I (Without Anaesthesia)
Description: The Schirmer test Type I (without anaesthesia) was performed to measure aqueous tear secretion prior to the instillation of any dilating or anaesthetic eye drops. The rounded bent end of a sterile strip was inserted into the lower conjunctival sac over the temporal one-third of the lower eyelid margin. After 5 minutes had elapsed, the Schimer's test strip was removed and the length of the tear absorption on the strip was measured (millimeters/5 minutes). The longer the wetted length, the healthier the status of the eye.
Time Frame: Visit 3 - Day 14±2, Visit 4 - Day 28±4, Visit 5 - Final visit/Follow up - Day 31- 41
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/5min
Arm/Group | Lubricin PP | Sodium Hyaluronate PP
Number analyzed (Participants) | 24 | 27
mm/5min
  Day 14±2 - Study eye | 0.7 (2.4) | 1.0 (2.8)
  Day 14±2 - Non study eye | 0.9 (2.5) | 1.5 (3.1)
  Day 28±4 - Study eye | 1.2 (3.6) | 0.9 (2.5)
  Day 28±4 - Non study eye | 1.1 (3.2) | 1.5 (2.6)
  Day 31-41 - Study eye | 0.5 (1.9) | 0.3 (2.0)
  Day 31-41 - Non study eye | 0.4 (1.6) | 0.7 (2.3)
Statistical Analysis 1: Comparison: Lubricin PP vs Sodium Hyaluronate PP; Study eye analytic statistic is presented.The Statistical Analysis section reports results from a repeated measures ANOVA, which analyzes changes from baseline (Visit 2 - Day 1) across all time points in a single unified analysis. This approach provides one overall comparison value by incorporating all time points. Consequently, the reported value represents the global outcome, consistently with repeated measures ANOVA methodology; Test type: Superiority; p = 0.6248, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.62 to 1.02]

10. Secondary Outcome: Change From Baseline in Intraocular Pressure (IOP)
Description: The IOP (intraocular pressure) of the eye was determined by the balance between the amount of aqueous humor that the eye marked and ease with which it leaved the eye. IOP was performed using Goldmann applanation tonometry after the instillation of a topical anaesthetic. The Goldmann applanation tonometer measured the force necessary to flatten a corneal area of 3.06 mm diameter. At this diameter, the resistance of the cornea to flattening was counterbalanced by the capillary attraction of the tear film meniscus for the tonometer head. The IOP (in mm Hg) equals the flattening force (in grams) multiplied by 10. IOP was measured in both eyes after completion of all SLEs to avoid potential interference with the other evaluations. Both eyes were tested. Normal eye pressure was between 10 to 21 mmHg. High ocular pressure was greater than 21 mmHg.
Time Frame: Visit 3 - Day 14±2, Visit 4 - Day 28±4, Visit 5 - Final visit/Follow up - Day 31- 41
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lubricin PP | Sodium Hyaluronate PP
Number analyzed (Participants) | 24 | 27
mmHg
  Day 14±2 - Study eye | 0.7 (1.9) | -0.6 (2.1)
  Day 14±2 - Non study eye | -0.4 (2.1) | -0.2 (1.9)
  Day 28±4 - Study eye | -0.2 (1.8) | -0.4 (2.5)
  Day 28±4 - Non study eye | -0.3 (1.7) | 0.1 (2.6)
  Day 31-41 - Study eye | -0.8 (2.6) | -0.9 (2.5)
  Day 31-41 - Non study eye | -0.5 (2.5) | -0.2 (2.6)
Statistical Analysis 1: Comparison: Lubricin PP vs Sodium Hyaluronate PP; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.6153, ANOVA; The analysis of variance included as sources of variability treatment, site and baseline tolerability score; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.82 to 0.49]

ADVERSE EVENTS:
Time Frame: AEs were assessed throughout the clinical investigation (V1 at Day -14 - -8; V2 at Day 1; V3 at Day 14 ± 2; V4 at Day 28 ± 4) up to final visit, at day 31- 41 (V5).
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product, which did not necessarily have a causal relationship with the treatment. An AE could be any unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease temporally associated with the use of a medicinal product. The adverse Events were reported at the patient level at both eyes.
Groups:
- Sodium Hyaluronate SAF: Sodium hyaluronate 0.13% eye drops. The comparator, as well as the test investigational device, was instilled i.d.(four times a day), one drop into each eye for 28±4 days. After the end of the treatment period, all the subjects used 0.13%Sodium hyaluronate eye drops q.i.d. for the following 7-9 days.
  Before the start of the treatment (run-in period of 7 days), the subjects were allowed to use NaCl 0.9% ocular solution q.i.d.
  Sodium Hyaluronate: Sodium hyaluronate 0.13% eye drops
Arm/Group | Lubricin SAF | Sodium Hyaluronate SAF
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/29
Other Adverse Events (participants affected / at risk) | 1/27 | 2/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lubricin SAF (N=27) | Sodium Hyaluronate SAF (N=29)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (4)
Eye oedema (Eye disorders) | 1 (1) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No